CLINICAL TRIAL: NCT03155698
Title: Treatment of Acral Vitiligo : Narrowband Ultraviolet-B and Microneedling With and Without Platelet Rich Plasma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lamia Ahmed, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOAV
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be randomized to treatment with microneedling by using dermapen every two weeks while the contralateral side of the body will be treated by microneedling plus topical PRP every two weeks .Then both sides of the body will receive narrowband UVB twice weekly for 6 month,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- microneedling,NB-UVB with & without PRP (Experimental): Each participant will be compared with one side of the body to the other side
  Intervention:
  * Combination Product: microneedling and Platelet rich plasma.
  * radiation : NB-UVB phototherapy
  Interventions: Combination Product: microneedling and Platelet rich plasma; Radiation: NB-UVB phototherapy

INTERVENTIONS:
Combination Product: microneedling and Platelet rich plasma — Patient's skin is first cleaned with ethyl alcohol. Topical anaesthetic cream is then applied to skin for 30 min. Once anaesthesias is fully developed, Dermapen will be applied on the lesional skin in four direction, vertical, horizontal and the two diagonal until pin point bleeding occur which will be gently massaged.
  * After ten minutes the prepared platelet rich plasma will be applied topically and after about 2 minutes. Occlusive dressing will be done and kept for 1 day then the patient will use topical antibiotic. The procedure will be repeated every 15 days.
  Other Names: dermapen+ topical PRP
Radiation: NB-UVB phototherapy — All patients will receive NB-UVB twice weekly for maximum 6 months, starting with a dose of 0.21 J/cm² independent of skin type and increased by 20% every session until we reach the minimal erythema dose

SUMMARY:
Vitiligo is a relatively common acquired chronic disorder of pigmentation characterized by the development of white macules on the skin due to loss of epidermal melanocytes .Affecting approximately 0.5%-2% of general population worldwide, without predilection for sex or race.

DETAILED DESCRIPTION:
Lesions may occur in a localized or generalized distribution and may coalesce into large, depigmented areas. Given the contrast between the white areas and normal skin, the disease is most disfiguring in darker skin types and has a profound impact on the quality of life of both children and adults. Generalized vitiligo is the most common clinical presentation and often involves the face and acral regions. The acral and joint areas are common sites of occurrence of vitiliginous lesions, because they are areas subjected to repeated trauma or irritation . The acral lesions are more visible and cosmetically important than lesions at many other sites, causing greater psychosocial distress Acral lesions are usually more resistant to medical management . Several reasons have been put forward, including relatively low melanocyte density; minimal density of hair follicles, which are a melanocyte reservoir; and a greater chance of repeated friction or trauma, which can induce koebnerization. Both acral and joint lesions also tend to be resistant to surgical management . The narrow band-ultraviolet B phototherapy is considered to be a very important modality in vitiligo treatment since its first use in 1997. It was proved to be of higher efficacy, better tolerated, and superior to the other lines of treatment . The prolonged duration of narrow band-ultraviolet B therapy is the main reason for noncompliance, distance to be traveled and monetary, and time loss in attending the hospital at least twice a week for prolonged time were cited as the second common cause for attrition. This clearly increases the need for combined therapy with narrow band-ultraviolet B (NB-UVB) to shorten the duration.

Combined treatments have been found to be superior to monotherapies regarding efficacy, early response and safety, especially in difficult to treat areas and refractory cases .

Platelet-rich plasma (PRP) is an autologous preparation of platelets in concentrated plasma.

Various growth factors, including platelet-derived growth factor, transforming growth factor, vascular endothelial growth factor, and insulin-like growth factor, are secreted from α-granules of concentrated platelets activated by aggregation inducers .

The beneficial effect of platelet rich plasma in vitiligo could be suggested through these growth factors which stimulate keratinocytes and fibroblasts proliferation with subsequent improvement of their interaction with melanocytes leading to the stabilization of melanocytes, it was also found that platelet rich plasma treatment induced accelerated proliferation and migration of fibroblasts through up-regulation of cyclin E and Cyclin- dependent kinase 4, which is important in cell migration and proliferation . Skin micro needling is a technique predominantly used to improve the appearance of cutaneous scarring and photo damage, fine needles puncture the skin, resulting in increased dermal elastin and collagen, collagen remodeling, and thickening of the epidermis and dermis . Additionally, skin needling creates small channels, which increase the absorption of topically applied preparations which has been used in various dermatological treatments.

.Aim of the work:

1. To determine efficacy and safety of automated microneedling + topical platelet rich plasma in combination with narrowband- ultraviolet B in treatment of resistant acral vitiligo.
2. To compare the efficacy of automated microneedling + topical Platelet rich plasma in combination with narrowband ultraviolet B versus automated microneedling and narrowband ultraviolet B only in treatment of resistant acral vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Patients with bilateral and symmetrical vitiligo acral in distribution.
* Lesions stable for at least three months.
* Patients receiving topical treatment will be required to undergo two weeks washout period.
* Patients receiving systemic treatment will be required to undergo 1 month washout period.
* Patients who were unresponsive to medical treatment or photo therapy.
* No sex predilection

Exclusion Criteria:

* Haemoglobin< 10 g/dl.
* Platelet count < 105 /UL.
* Patients with active infection.
* Reported histories of koebnerization.
* History of keloid formation or hypertrophic scars.
* Pregnant or lactating females.
* Bleeding tendency.
* Patients with chronic liver diseases.
* Patients using systemic chemotherapy, anti-coagulation therapy and antiplatelet agents.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
VASI score-Vitiligo Area and Severity Index | within 6 months
  Vitiligo Area and Severity Index (VASI) One hand unit, which encompasses the palm plus the volar surface of all the digits, is approximately 1% of the total body surface area and is used to estimate the baseline percentage of vitiligo involvement in each body region. The body is divided into five separate and mutually exclusive regions: hands, upper extremities (excluding hands), trunk, lower extremities (excluding feet), and feet. The axillary region is included with the upper extremities while the buttocks and inguinal areas are included with the lower extremities. The extent of residual depigmentation is expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%. At 100% depigmentation, no pigment is present; at 90%, specks of pigment are present; at 75%, the depigmented area exceeds the pigmented area; at 50%, the depigmented and pigmented areas are equal; at 25%, the pigmented area exceeds the depigmented area; at 10%, only specks of depigmentation

SECONDARY OUTCOMES:
scoring system of repigmentation | assessed 6 months following application of intervention
  * G0, < 25% repigmentation (poor)
  * G1, 25-50% repigmentation (fair)
  * G2, 50-75% repigmentation (good)
  * G3 > 75% repigmentation (excellent).
Patients satisfaction | within 6months
  The patient overall satisfaction will be assessed according to Overall satisfaction:
  1. dissatisfied
  2. neutral
  3. somewhat satisfied
  4. moderately satisfied
  5. very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa Ahmad Abd El-khalek, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ezzedine K, Eleftheriadou V, Whitton M, van Geel N. Vitiligo. Lancet. 2015 Jul 4;386(9988):74-84. doi: 10.1016/S0140-6736(14)60763-7. Epub 2015 Jan 15. PMID 25596811
- [Result] Kruger C, Schallreuter KU. Stigmatisation, Avoidance Behaviour and Difficulties in Coping are Common Among Adult Patients with Vitiligo. Acta Derm Venereol. 2015 May;95(5):553-8. doi: 10.2340/00015555-1981. PMID 25269389
- [Result] Olsson MJ, Juhlin L. Long-term follow-up of leucoderma patients treated with transplants of autologous cultured melanocytes, ultrathin epidermal sheets and basal cell layer suspension. Br J Dermatol. 2002 Nov;147(5):893-904. doi: 10.1046/j.1365-2133.2002.04837.x. PMID 12410698
- [Result] Holla AP, Parsad D. Vitiligo surgery: its evolution as a definite treatment in the stable vitiligo. G Ital Dermatol Venereol. 2010 Feb;145(1):79-88. PMID 20197747
- [Result] Westerhof W, Nieuweboer-Krobotova L. Treatment of vitiligo with UV-B radiation vs topical psoralen plus UV-A. Arch Dermatol. 1997 Dec;133(12):1525-8. PMID 9420536
- [Result] Kandaswamy S, Akhtar N, Ravindran S, Prabhu S, Shenoi SD. Phototherapy in Vitiligo: Assessing the Compliance, Response and Patient's Perception about Disease and Treatment. Indian J Dermatol. 2013 Jul;58(4):325. doi: 10.4103/0019-5154.113944. PMID 23919018
- [Result] Kaux JF, Le Goff C, Seidel L, Peters P, Gothot A, Albert A, Crielaard JM. [Comparative study of five techniques of preparation of platelet-rich plasma]. Pathol Biol (Paris). 2011 Jun;59(3):157-60. doi: 10.1016/j.patbio.2009.04.007. Epub 2009 May 28. French. PMID 19481375
- [Result] Aust MC, Reimers K, Kaplan HM, Stahl F, Repenning C, Scheper T, Jahn S, Schwaiger N, Ipaktchi R, Redeker J, Altintas MA, Vogt PM. Percutaneous collagen induction-regeneration in place of cicatrisation? J Plast Reconstr Aesthet Surg. 2011 Jan;64(1):97-107. doi: 10.1016/j.bjps.2010.03.038. Epub 2010 Apr 21. PMID 20413357
- [Result] Fabbrocini G, De Vita V, Izzo R, Monfrecola G. The use of skin needling for the delivery of a eutectic mixture of local anesthetics. G Ital Dermatol Venereol. 2014 Oct;149(5):581-5. PMID 25213385
- [Result] Gonshor A. Technique for producing platelet-rich plasma and platelet concentrate: background and process. Int J Periodontics Restorative Dent. 2002 Dec;22(6):547-57. PMID 12516826